CLINICAL TRIAL: NCT03613766
Title: A Supervised Exercise Program Reduces Fat Mass and Cardiovascular Risk Factors in Patients Awaiting Bariatric Surgery
Brief Title: Physical Activity Program Before Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Manuel Moya, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016.234.E.OEP
Record Dates: First submitted 2018-07-09; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Bariatric Surgery Candidate; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Two groups (experimental and control). Chronological order of recruitment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity program (Experimental): Before 3 to 6 months before the expected date of surgery, the experimental group, performed a 12-week monitored and supervised concurrent exercise program. Before and after of this period, body composition, anthropometric measures, physical fitness, cardiovascular risk, blood samples, Basal Metabolic Rate and health-related quality of life were measured in a laboratory under controlled conditions.
  Interventions: Other: Physical activity program
- Habitual care prescription (No Intervention): Before 3 to 6 months before the expected date of surgery, the control group, followed the habitual care prescriptions until the surgery

INTERVENTIONS:
Other: Physical activity program
  Arms: Physical activity program

SUMMARY:
Background: Weight reduction, especially of visceral fat in patients awaiting bariatric surgery (BS), may facilitate the surgical process, and reduce postoperative complications. Normally, to achieve weight reductions a nutritional treatment is prescribed, but the effects of exercise on these patients have been little studied.

Objectives: To know the effects of an exercise program on body composition and cardiovascular risk factors in patients awaiting BS.

Methods: Twenty-three patients awaiting BS were divided into two groups: a) an experimental group (EG, n = 12); b) a control group (CG, n = 11). Both groups received the usual care prior to surgery, but the EG also performed a 12-week exercise program in which endurance and resistance training were combined. Body composition, anthropometric measures, cardiovascular risk factors, physical fitness, basal metabolic rate and quality of life were assessed at baseline and at the end of the study.

DETAILED DESCRIPTION:
Patients included in the presurgical protocol for BS at two University Hospitals were recruited while awaiting surgery. Each patient participated in an initial interview, during which all the aspects of the program were carefully explained, and a written informed consent was obtained. After that, the individual's medical history was checked looking for the presence of the following exclusion criteria: a) cardiovascular diseases; b) severe functional limitations; c) chronic respiratory diseases; or d) being undergoing another exercise program at the time of the study. Finally, twenty-three participants were diachronically enrolled in the intervention at 3 to 6 months before the expected date of surgery. The patients were assigned to the experimental group (EG) or to the control group (CG) in chronological order of recruitment: the first 12 patients were included in the EG, and the other 11 patients in the CG. The study protocol was approved by the local ethics committee and conformed to the Declaration of Helsinki.

Both groups followed the usual presurgical care of their respective hospitals (psychological and nutritional counseling). In addition, the EG performed a 12-week monitored and supervised CEP, while the CG only received advice to follow an active lifestyle. Both groups were assessed at the start (T1) and the end of the study, after 12 weeks (T2). At each assessment session, body composition, anthropometric measures, physical fitness, cardiovascular risk (CVR) and CVR factors, basal metabolic rate (BMR) and health-related quality of life were measured in a laboratory under controlled conditions (temperature 22-24º; relative air humidity 45-60%). Blood samples from each patient were taken and analyzed in their respective hospitals at the same timepoints.

Concurrent exercise program (CEP) The CEP was divided into three 4-week blocks, for a total duration of 12 weeks. In the first-block endurance training (ET) (performed on a cycle-ergometer, arm-ergometer, elliptical and treadmill) and resistance training (RT) (performed in resistance machines for 5 muscle groups: hamstrings, pectorals, quadriceps, latissimus dorsi, and gastrocnemius) were combined in the same session. During the second-block, patients performed 3 sessions per week. One day, only ET was performed. In the other 2 sessions, patients performed a High Intensity Interval Training (HIIT) on a cycle ergometer or an arm-ergometer followed by 7 resistance exercises (biceps and triceps brachii were added to the previous 5 major muscle groups trained).

In the third-block, patients trained 4 days a week. Two days a week, HIIT and RT were combined in the same session. RT was performed after HIIT. It consisted in training 4 different major muscle groups in each session (pectorals, quadriceps, biceps, and hamstrings in the first session, and latissimus dorsi, triceps, gastrocnemius and deltoids in the second session). In the other two sessions, only ET was carried out. In all the blocks, 2 days a week of flexibility training were carried out.

The intensity of the ET was monitored using a heart rate (HR) monitor (FT40, Polar, Finland), while the intensity of the RT was determined by percentages of 1 maximum repetition, which was estimated using the Brzycki formula.

The HIIT performed consisted of a 5-minute warm-up, followed by the main part of 20 minutes with bouts of 30 seconds at high intensity (60-80% VO2peak) and 30 seconds of active recovery (40% VO2peak), for a total of 10 minutes of training at high intensity. Once the main part was finished, 3 minutes of cool-down at 40% VO2peak were performed. The rate of perceived exertion (RPE) was taken of each session using the CR-10 Borg's scale in order to control the progression of training loads.

Anthropometry and body composition. These measures were performed between 7:30 and 8:30 A.M., after 10-12 hours overnight fast, with an empty bladder. Exercise was forbidden in the 72 hours before the test, as well as the consumption of caffeine or alcohol in the 24 hours before the test. Waist and hip circumference and height were measured using the ISAK (International Society for the Advancement of Kinanthropometry) protocol. Total weight and body composition were measured by bioimpedance analysis (Tanita BC-420MA, Tanita, Tokyo, Japan). Body mass index was calculated, and expressed as kg·m-2.

Cardiorespiratory fitness. A protocol in cycle ergometer (Technogym Bike Med, Technogym, Gambettola, Italy) adapted Achten was used to determine the peak oxygen uptake (VO2peak) using an Oxycon Pro gas analysis system (Jaeger, Friedberg, Germany). This protocol consisted of two phases. In the first phase, patients performed a 4 -minutes warm-up at 40 watts (W), followed by increases of 20 W every 3 minutes, maintaining a cadence of 60 rotations per minute (RPM), until the respiratory exchange ratio (RER) reached 1.0. At this point the second phase started, which consisted of increments of 20 w each minute, maintaining a cadence between 70-80 RPM, until volitional fatigue. The average of the highest 30 seconds of VO2 was used to calculate VO2peak. The VO2peak was expressed in absolute values (VO2peak abs) and normalized to total body weight (VO2peak/BW) and fat- free mass (VO2peak/FFM). Subjects with musculoskeletal disorders on the leg performed the same test in an arm-ergometer but initiated at 20W with increases of 10 W (Technogym, Excite®+Top MD Inclusive).

Muscle strength Dynamic and isometric strength of the quadriceps, hamstrings, biceps and triceps brachii were assessed using an isokinetic dynamometer (Biodex System 4; Biodex Medical Systems, New York, USA). First, patients performed a 5-minute warm-up on a cycle ergometer at an intensity of 60% of individual HRmax. Next, participants were stabilized on the dynamometer chair (seat back angle ~ 85º) with two shoulder straps and a thigh strap. The anatomical axis of rotation was aligned to the dynamometer axis to allow movement in the sagittal plane for the knee and in the transversal plane for the elbow. For each limb, 3 unipodal tests were performed, 1 isokinetic test and 2 isometric tests. A two-minutes rest was conducted between tests and 3 minutes between limbs.

Dynamic strength measurement (MDS): Participants performed 4 sets of 4 concentric contractions (flexion-extension) of the upper (elbow) and lower body (knee), at an angular speed of 60º/s, with 90 s rest between repetitions. The knee and elbow motion ranges were within 105° to 10° and within 160° to 60°, respectively. The first series was a submaximal familiarization trial. In the following three sets, participants were verbally encouraged to perform and maintain maximal effort in every contraction. The peak torque (N·m) of each set was analyzed and the average of the last three sets was calculated. Additionally, the peak torque was normalized to the individual's body weight (MDSBW) and relative to FFM (MDSFFM).

Isometric strength measurement (MIS): Participants completed a submaximal repetition followed by 3 maximum voluntary contraction (15 s rest between repetitions), during which they were verbally encouraged to perform a maximal effort for 5 s, following the recommendations of previous research .(40). The angles used for assessing quadriceps and hamstrings were of 105º and 75º, respectively, and triceps and biceps brachii were of 75º and 120º, respectively. As there was one set per exercise, the peak torque (N·m) was analyzed and normalized to the body weight (MISBW) and individual's FFM (MISFFM).

Basal metabolic rate BMR was calculated by indirect calorimetry, using an Oxycon Pro gas analysis system (Jaeger, Friedberg, Germany). The patients were 30 minutes in supine position in a comfortable bed. To perform the analysis, only the data from the last 10 minutes of the assessment were used. BMR was determined according to the Weir formula and, was normalized to BW (BMRBW) and to FFM (BMRFFM). BMR was measured at the same times and under the same ambient conditions that anthropometry and body composition measurements.

Cardiovascular risk factors. Blood samples were taken at the University Hospitals, after 12 hours overnight fast. Patients were instructed not to perform exercise 48 hours before the test. Standard methods were used to measure total cholesterol (TC), HDL cholesterol (HDL-C), glucose, HbA1C, and triglycerides (TG). Friedwald equation was used for calculating LDL cholesterol (LDL-C) (42). Blood pressure was measured according to established recommendations, using a digital sphygmomanometer (Microlife WatchBP Home, Heerbrugg, Switzerland).

Framingham cardiac risk score adapted to the Spanish context was used to calculate CVR. This formula, uses the TC, HDL-C, blood pressure values, sex, age, diabetic and/or smoking status, to calculate the 10-year coronary risk. In some subjects of the CG, this formula could not be applied, since they were less than 35 years old, thus, CVR was also determined by the waist-to-hip ratio (WHpR) and by the waist-to-height ratio (WHtR).

Health-related quality of life. The Short Form Health Survey 36 (SF-36) in its version adapted to the Spanish context was used to determine health related to the life quality of the patients. Physical and mental health are measured by 8 scales, the scores of which are transformed to values between 0-100 points, indicating the highest scores a better function. These 8 scales are grouped into two summary components (physical and mental) (49), which were calculated according to the reference values of the Spanish population (50), with a mean of 50 and standard deviation of 10.

ELIGIBILITY:
Inclusion Criteria:

1. Be on the surgery waiting list.
2. Follow the doctor's usual health prescriptions

Exclusion Criteria:

1. cardiovascular diseases
2. severe functional limitations
3. chronic respiratory diseases
4. being undergoing another exercise program at the time of the study

Ages: 35 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Body Composition at 3 months | Baseline and 3 months, between 7:30 AM and 8:30 AM.
  Body mass index (BMI) was calculated according to the formula: total weight in kilograms divided by squared height in meters (kg·m-2). Participants performed the assessment with an empty bladder. Bioimpedance analysis (Tanita BC-420MA, Tanita, Tokyo, Japan) was used to establish body weight and body composition.
Change from Baseline Cardiorespiratory Fitness at 3 months | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  A protocol in cycle ergometer (Technogym Bike Med, Technogym, Gambettola, Italy) adapted Achten was used to determine the peak oxygen uptake (VO2peak) using an Oxycon Pro gas analysis system (Jaeger, Friedberg, Germany). This protocol consisted of two phases. In the first phase, patients performed a 4-minutes warm-up at 40 watts (W), followed by increases of 20 W every 3 minutes, maintaining a cadence of 60 rotations per minute (RPM), until the respiratory exchange ratio (RER) reached 1.0. At this point the second phase started, which consisted of increments of 20 w each minute, maintaining a cadence between 70-80 RPM, until volitional fatigue. The average of the highest 30 seconds of VO2 was used to calculate VO2peak. The VO2peak was expressed in absolute values (VO2peak abs) and normalized to total body weight (VO2peak/BW) and fat- free mass (VO2peak/FFM)
Change from Baseline Muscle strength at 3 months. Dynamic strength measurement | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  Dynamic and isometric strength of the quadriceps, hamstrings, biceps and triceps brachii were assessed using an isokinetic dynamometer (Biodex System 4; Biodex Medical Systems, New York, USA). Participants performed 4 sets of 4 concentric contractions (flexion-extension) of the upper (elbow) and lower body (knee), at an angular speed of 60º/s, with 90 s rest between repetitions. The knee and elbow motion ranges were within 105° to 10° and within 160° to 60°, respectively. The first series was a submaximal familiarization trial. In the following three sets, participants were verbally encouraged to perform and maintain maximal effort in every contraction. The peak torque (N·m) of each set was analyzed and the average of the last three sets was calculated. Additionally, the peak torque was normalized to the individual's body weight (MDSBW) and relative to FFM (MDSFFM)
Change from Baseline Muscle strength at 3 months. Isometric strength measurement | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  Dynamic and isometric strength of the quadriceps, hamstrings, biceps and triceps brachii were assessed using an isokinetic dynamometer (Biodex System 4; Biodex Medical Systems, New York, USA). Participants completed a submaximal repetition followed by 3 maximum voluntary contraction (15 s rest between repetitions), during which they were verbally encouraged to perform a maximal effort for 5 s, following the recommendations of previous research. The angles used for assessing quadriceps and hamstrings were of 105º and 75º, respectively, and triceps and biceps brachii were of 75º and 120º, respectively. As there was one set per exercise, the peak torque (N·m) was analyzed and normalized to the body weight (MISBW) and individual's FFM (MISFFM).
Change from Baseline Cardiovascular risk factors at 3 months. | Baseline and 3 months, in a different day of the other tests, between 8:00 AM and 9:00 AM.
  Blood samples were taken at the University Hospitals, after 12 hours overnight fast. Patients were instructed not to perform exercise 48 hours before the test. Standard methods were used to measure total cholesterol (TC), HDL cholesterol (HDL-C), glucose, HbA1C, and triglycerides (TG). Friedwald equation was used for calculating LDL cholesterol (LDL-C). Blood pressure was measured according to established recommendations, using a digital sphygmomanometer (Microlife WatchBP Home, Heerbrugg, Switzerland).
  Framingham cardiac risk score adapted to the Spanish context was used to calculate CVR. This formula, uses the TC, HDL-C, blood pressure values, sex, age, diabetic and/or smoking status, to calculate the 10-year coronary risk. In some subjects of the CG, this formula could not be applied, since they were less than 35 years old, thus, CVR was also determined by the waist-to-hip ratio (WHpR) (45) and by the waist-to-height ratio (WHtR)
Change from Baseline waist and hip circumference at 3 months | Baseline and 3 months, between 7:30 AM and 8:30 AM.
  The ISAK (International Society for the Advancement of Kinanthropometry) protocol was used to assess waist and hip circumference.

SECONDARY OUTCOMES:
Change from Baseline Basal metabolic rate at 3 months | Baseline and 3 months, in a different day of the other tests, between 8:00 AM and 9:00 AM.
  It was calculated by indirect calorimetry, using an Oxycon Pro gas analysis system (Jaeger, Friedberg, Germany). The patients were 30 minutes in supine position in a comfortable bed. To perform the analysis, only the data from the last 10 minutes of the assessment were used. BMR was determined according to the Weir formula and was normalized to BW (BMRBW) and to FFM (BMRFFM).
  BMR was measured at the same times and under the same ambient conditions that anthropometry and body composition measurements.
Change from Baseline Health-related quality of life at 3 months | Baseline and 3 months, between 8:00 AM and 9:00 AM.
  The Short Form Health Survey 36 (SF-36) in its version adapted to the Spanish context was used to determine health related to the life quality of the patients. Physical and mental health are measured by 8 scales, the scores of which are transformed to values between 0-100 points, indicating the highest scores a better function. These 8 scales are grouped into two summary components (physical and mental), which were calculated according to the reference values of the Spanish population, with a mean of 50 and standard deviation of 10

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marc-Hernandez A, Ruiz-Tovar J, Aracil A, Guillen S, Moya-Ramon M. Impact of Exercise on Body Composition and Cardiometabolic Risk Factors in Patients Awaiting Bariatric Surgery. Obes Surg. 2019 Dec;29(12):3891-3900. doi: 10.1007/s11695-019-04088-9. PMID 31313237